CLINICAL TRIAL: NCT05797779
Title: Molecular Characterization of Induced Neuronal Cells Derived From Fibroblasts of Patients With Parkinson's Disease
Brief Title: Molecular Characterization of Induced Neuronal Cells in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3482
Record Dates: First submitted 2023-02-28; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin biopsy (Experimental)
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Procedure: Skin biopsy — Punch biopsy of the skin

SUMMARY:
To describe the molecular, electrophysiological and morphological expression profile of dopaminergic neurons derived from fibroblasts of patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years or older
2. Patients with Parkinson's disease, according to the most recent diagnostic criteria
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study

Exclusion Criteria:

1. Patients affected by drug-induced parkinsonism or atypical parkinsonian disorders
2. Patients with neurological diseases other than Parkinson's disease
3. Inability to sign an informed consent
4. Severe psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological characterization of dopaminergic neurons derived from patients with Parkinson's disease. | Baseline
  To evaluate the firing frequency in the dopaminergic neurons derived from fibroblasts of patients with Parkinson's disease.
Biochemical characterization of dopaminergic neurons derived from patients with Parkinson's disease. | Baseline
  To determine the amount of dopamine released from differentiated neurons derived from fibroblasts of patients with Parkinson's disease.
α-synuclein misfolding in dopaminergic neurons derived from patients with Parkinson's disease. | Baseline
  To document the presence of abnormal accumulation of misfolded alpha-synuclein in the dopaminergic neurons derived from fibroblasts of patients with Parkinson's disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Flavia Torlizzi, Roma, Italy